CLINICAL TRIAL: NCT03322722
Title: Implementation of a Tool on Alimentary Empowerment in New-born Baby
Status: Completed | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: LAVOILACTEE
Record Dates: First submitted 2017-10-16; First posted 2017-10-26 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Neonatal Feeding Disorder

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The alimentation of the premature newborn children is one of main thing concerning of nurses and pediatricians in neonatology. The absence of common tool of evaluation of the children cause a great discrepancy in prescriptions and the practices of the nursing.The aim of this study is to estimate the improvement of the food empowerment of the premature newborn children after the introduction of a help tool at the food progress which allows to fit the prescription of food(supply) to the capacities of the newborn child.

DETAILED DESCRIPTION:
If the importance of feeding premature newborns is a central concern during their management, the absence of an evaluation tool leads to a great disparity in their implementation (particularly marked by at regular times by the care teams), which can eventually lead to oral disorders. The possibility of an assessment of the newborn's skills could allow a homogenization of therapeutic proposals and thus a potentially faster progression of dietary independence of the newborn. This method could also encourage parental involvement in feeding care. The objective of the study is to evaluate the impact of a tool to help food progression on food autonomy.

ELIGIBILITY:
Inclusion Criteria:

* born before 37 weeks of pregnancy
* hospitalized in GHPSJ neonatology
* Predictable duration of hospitalization of at least 7 days

Exclusion Criteria:

* parents not speaking french language
* new borm with complication du to his prematurity

Ages: 1 Day to 5 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: every baby born before 37 weeks of pregnancy between january 2017 and end of march 2017
Sampling Method: Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2016-10-14 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2022-12-07 (Actual)

PRIMARY OUTCOMES:
Age of prematurity of the newborn child | delivery date
  It's an estimation between the real age of the premature baby (i.e number of weeks of pregnancy) and the normal date of delivery.

CONTACTS AND LOCATIONS:
Overall Officials: SUILS Hélène, MD, Principal Investigator — Fondation Hôpital Saint-Joseph
Locations (1):
- Groupe Hospitalier Paris Saint Joseph, Paris, Île-de-France Region, France